CLINICAL TRIAL: NCT06577558
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of SR1375 in Hospitalized Adult Patients With Community-acquired Pneumonia
Brief Title: Efficacy and Safety of SR1375 in Adult Patients With CAP
Acronym: CAP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SR1375-204
Record Dates: First submitted 2024-08-19; First posted 2024-08-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Community-acquired Pneumonia
Keywords: Community acquired Pneumonia; SR1375
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SR1375 capsule 3mg (Experimental): SR1375 capsule 3mg quaque die(QD) orally with CAP regular treatments for 8 weeks
  Interventions: Drug: SR1375 capsule 3mg+regular treatments
- SR1375 capsule 1mg (Experimental): SR1375 capsule 1mg QD orally with CAP regular treatments for 8 weeks
  Interventions: Drug: SR1375 capsule 1mg+regular treatments
- SR1375 capsule 0.3mg (Experimental): SR1375 capsule 0.3mg QD orally with CAP regular treatments for 8 weeks
  Interventions: Drug: SR1375 capsule 0.3mg+regular treatments
- placebo capsule (Placebo Comparator): Placebo capsule QD orally with CAP regular treatments for 8 weeks
  Interventions: Drug: Placebo capsule+regular treatments

INTERVENTIONS:
Drug: SR1375 capsule 3mg+regular treatments — SR1375 capsule 3mg QD orally+CAP regular treatments
  Other Names: SR1375 capsule high dose+regular treatments
  Arms: SR1375 capsule 3mg
Drug: SR1375 capsule 1mg+regular treatments — SR1375 capsule 1mg QD orally+CAP regular treatments
  Other Names: SR1375 capsule medium dose+regular treatments
  Arms: SR1375 capsule 1mg
Drug: SR1375 capsule 0.3mg+regular treatments — SR1375 capsule 0.3mg QD orally+CAP regular treatments
  Other Names: SR1375 capsule low dose+regular treatments
  Arms: SR1375 capsule 0.3mg
Drug: Placebo capsule+regular treatments — Placebo capsule QD orally+CAP regular treatments
  Arms: placebo capsule

SUMMARY:
This is a phase 2 study to evaluate the efficacy and safety of SR1375 in hospitalized adult patients with CAP. Patients will receive SR1375 or placebo for 8 weeks. The study duration for each patient is up to 10 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind and placebo-controlled phase 2 study comparing SR1375 with placebo in adult patients with CAP. It consists of a screening period, a double-blind treatment period, and a post-treatment safety follow-up period. Baseline NIAID-OS 8-point scale score will be checked for eligibility. Around 240 eligible subjects will be recruited and randomized into four arms at 1:1:1:1 ratio to receive SR1375 0.3mg, SR1375 1mg, SR1375 3mg or placebo orally daily for 56 days. Subjects, investigators, all clinical study site staffs, and the Sponsor will remain blinded to treatment assignment during the study. Subjects will receive regular treatments as per his/her condition by investigator. After completion of double-blind treatment period, subjects will continue to complete the safety follow-up for 14 days.

ELIGIBILITY:
Key Inclusion Criteria:

* The subject or their legally acceptable representative (LAR) has voluntarily signed the informed consent form (ICF) prior to any study-related procedures, and the subject is willing and able to comply with all study requirements, restrictions, and procedures. If consent is provided by an LAR for a subject with limited or no capacity to consent, re-consenting may be performed if the subject regains capacity.
* Aged 18 to 85 years.
* Diagnosis of CAP
* Prior to screening, the subject has been receiving standard-of-care treatment for pneumonia in a medical institution, including at least 3 days of intravenous (IV) anti-infective therapy, with no clinical improvement.
* Chest CT showing multi-lobar infiltrates, and for subjects not receiving invasive mechanical ventilation, an oxygenation index (PaO2/FiO2 ratio) between 100 and 300 mmHg.
* Expected to require continued hospitalization for at least 7 days from the time of signing the ICF.
* Baseline NIAID-OS 8-point scale score of 5 points and transcutaneous oxygen saturation ≤ 93% without oxygen inhalation, 6 points or 7points. (5 points refer to hospitalization with oxygen therapy; 6 points refer to hospitalization with high flow oxygen therapy or non-invasive mechanical ventilation. 7 points refer to hospitalization with invasive mechanical ventilation).High oxygen flow refers to ≥ 4 L/min.)
* With ≥ 1 high risk factors including chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, type 2 diabetes, chronic kidney disease, coronary heart disease, age ≥ 65 years, moderate obesity (body mass index>32.5kg/m2), etc.
* Participants of women of childbearing potential(WOCBP) and male participants with WOCBP partners must agree to use one or more effective contraceptive methods during the treatment period and until 90 days after the last administration.

Key Exclusion Criteria:

* Patients who are currently receiving or are expected to require ECMO treatment within 24 hours.
* Presence of active tuberculosis (TB) or severe asthma.
* History of unstable angina or acute myocardial infarction within 3 months prior to screening, or stroke within 4 weeks prior to screening.
* Received chemotherapy and/or immunotherapy for a malignant tumor within 4 weeks prior to randomization, or are planned to receive such treatment during the study period; presence of a hematological malignancy not in complete remission; or a lung tumor with concurrent obstructive pneumonia.
* Presence of any concomitant disease that is expected to result in death within 12 weeks after randomization.
* Prior use of JAK inhibitors (e.g., Baricitinib), interleukin receptor inhibitors (e.g., Tocilizumab), or any investigational drug in another clinical trial, where the last dose was administered less than 5 half-lives before the first dose of the study drug in this trial.
* ALT) or AST > 3 times the upper limit of normal (ULN).
* eGFR < 30 mL/min/1.73 m² (calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula); however, patients undergoing dialysis may be included upon the investigator's assessment of their suitability for the trial.
* Presence of clinically significant abnormalities on ECG that may seriously affect subject safety, e.g., QTcF > 480 ms.
* Female subjects who are pregnant, lactating, or have a positive serum β-HCG pregnancy test.
* Presence of any severe systemic disease or clinical condition that, in the investigator's judgment, makes the subject unsuitable for participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
National Institute of Allergy and Infectious Diseases-Outcome Study (NIAID-OS) 8-point scale score | Up to Day 28
  Change from baseline to Day 28 in NIAID-OS 8 scale score. NIAID-OS 8 scale ranges from 1 point (no hospitalization, no activity restrictions) to 8 points (death). The higher score means the worse outcome.

SECONDARY OUTCOMES:
Proportion of subjects ≥ 2 points improvement in National Institute of Allergy and Infectious Diseases-Outcome Study (NIAID-OS) 8-point scale score | Up to Day 28
  Subject proportion of ≥ 2 points improvement in NIAID-OS 8-point scale at Day 14 and Day 28
National Institute of Allergy and Infectious Diseases-Outcome Study (NIAID-OS) 8-point scale score | Up to Day 14
  Change from baseline to Day 7 and Day 14 in NIAID-OS 8 scale score. NIAID-OS 8 scale ranges from 1 point (no hospitalization, no activity restrictions) to 8 points(death)，the higher score means the worse outcome.
All-cause mortality rate | Up to Day 56
  The all-cause mortality rate at Day 28 and Day 56
Proportion of subjects with invasive mechanical ventilation, Extracorporeal Membrane Oxygenation(ECMO) or all-cause death. | Up to Day 56
  Subjects proportions with invasive mechanical ventilation, ECMO or all-cause death at Day 28 and Day 56.
Partial Pressure of Oxygen(PaO2)/Fraction of Inspiration Oxygen(FiO2) | Up to Day 28
  Change from baseline to Day 7 and Day 28 in PaO2/FiO2.
Proportion of subjects admitted in ICU or all-cause death | Up to Day 56
  Proportion of subjects admitted in ICU or all-cause death at Day 28 and Day 56
Proportion of subjects ≤ 2 points in NIAID-OS 8-point scale | Up to Day 56
  Proportion of subjects ≤ 2 points in NIAID-OS 8-point scale at Day 28 and Day 56
Survival days without invasive mechanical ventilation or ECMO | Up to Day 56
  Survival days without invasive mechanical ventilation or ECMO within 28 and 56 days.
Survival days without ICU admission | Up to Day 56
  Survival days without ICU admission within 28 and 56 days
Days of hospitalization | Up to Day 56
  Days of hospitalization within 28 and 56 days
All-cause readmission rate | Up to Day 56
  All-cause readmission rate within 56 days
Readmission rate due to pneumonia | Up to Day 56
  Readmission rate due to pneumonia within 56 days

OTHER OUTCOMES:
The item short from health survey (SF-36) score | Up to Day 56
  Change from baseline to Day 28 and Day 56 in SF-36 score. SF-36 scores range from 0 to 100 and the higher score means the better condition.
Adverse events and serious adverse events | Up to Day 70
  AE and SAE occurence and severity during the study
Pharmacokinetic (PK) parameter Cmax | Up to Day 56
  Maximum plasma concentration (Cmax) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
PK parameter Tmax | Up to Day 56
  Time to maximum concentration (Tmax) will be calculated by PhoenixWinNonlin software (V8.0 or higher) .
PK parameter AUC0-t | Up to Day 56
  Area under the concentration-time curve from 0 to the collection time t (AUC0-t) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
PK parameter t1/2 | Up to Day 56
  Half-Life (t1/2) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
PK parameter Vd/F | Up to Day 56
  Apparent volume of distribution (Vd/F) will be calculated by PhoenixWinNonlin software (V8.0 or higher).
Pharmacodynamic (PD) parameter lipoprotein associated phospholipase A2 (Lp-PLA2) activity | Up to Day 56
  PD parameter Lp-PLA2 activity will be tested in central laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Li, MD, Principal Investigator — West China Hospital
Locations (29):
- China (29):
  - Fuyang People's Hospital, Fuyang, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhangzhou Hospital, Zhangzhou, Fujian
  - Gaozhou People's Hospital, Gaozhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Yulin First People's Hospital, Yulin, Guangxi
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing Longnan Hospital, Daqing, Heilongjiang
  - Daqing People's Hospital, Daqing, Heilongjiang
  - Shangqiu People's Hospital, Shangqiu, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Yueyang Central Hospital, Yueyang, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Yanbian University Affiliated Hospital, Yanbian, Jilin
  - Dalian Central Hospital, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Weifang Second People's Hospital, Weifang, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - Lishui Central Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No